CLINICAL TRIAL: NCT04161833
Title: Use of an Alfa-lipoic, Methylsulfonylmethane and Bromelain Dietary Supplement (Opera®) for Aromatase Inhibitor-related Arthralgia Management (AIA)
Brief Title: Opera® for Aromatase Inhibitor-related Arthralgia Management (AIA)
Acronym: AIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Lorenzo Livi, Professor, Azienda Ospedaliero-Universitaria Careggi
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OPERA2
Record Dates: First submitted 2019-11-08; First posted 2019-11-13 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Breast Cancer; Hormone Receptor Positive Tumor; Arthralgia
Keywords: breast cancer; luminal tumor; anti-aromatase inhibitors; arthralgia; dietary supplement
MeSH Terms: conditions — Breast Neoplasms; Arthralgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OPERA (Experimental): Women receiving adjuvant aromates-inhibitor with arhtralgia grade ≥ 1 (CTACAE 4.03)
  Interventions: Dietary Supplement: OPERA

INTERVENTIONS:
Dietary Supplement: OPERA — All patients were required to take an OPERA® capsule (dietary supplement where α-lipoic acid, Boswellia Serrata, methylsulfonylmethane and bromelain are combined in a single capsule) once daily,from enrollment up to sixth months.

SUMMARY:
In this phase II, multicenter, self-controlled clinical trial, we will evaluate the safety and efficacy of OPERA® for treating anti-aromate inhibitors (AIs) induced arthralgia. The diagnosis of arthralgia will be based on the NCI-CTCAE v4.0 grade of ≥ 1 , A disorder characterized by a sensation of marked discomfort in a joint, mild pain (grade 1). Arthralgia will be assessed at the enrollment and every two months until the sixth month.

DETAILED DESCRIPTION:
Aromatase Inhibitors (AIs) are recommended for the adjuvant treatment of hormone receptor positive breast cancers in the post-menopausal population. Compared with Tamoxifen, third generation aromatase inhibitors have been shown to significantly improve disease free survival (DFS), and include the steroidal inhibitor exemestane, and the nonsteroidal inhibitors, anastrozole and letrozole. Although the AIs are associated with fewer thromboembolic events and endometrial abnormalities than is tamoxifen, approximately 25% of postmenopausal women on AI report arthralgia, skeletal, and muscle pain. The multicentre double-blind placebo-controlled ma.17 trial by the National Cancer Institute of Canada Clinical Trials Group revealed marked increases in arthralgia (25% vs. 21%) and myalgia (15% vs. 12%) in patients on letrozole as compared with those on placebo. The Intergroup Exemestane Study shown a link between arthralgia and the ai exemestane (5.4% exemestane vs. 3.6% tamoxifen).The Arimidex, Tamoxifen Alone or in Combination (atac) trial, after 68 months' median follow-up, showed that the incidence of arthralgia was significantly higher in the anastrozole group than in the tamoxifen group [1100 of 3092 (35.6%) vs. 911 of 3094 (29.4%) patients]. Currently, evidences of drugs efficacy to reduce these side effects are sparse.OPERA® (GAMFARMA srl, Milan, Italy) is a new dietary supplement where α-Lipoic acid (240mg), BS (40mg), MSM (200mg) and Bromelain (20mg) are combined together in a single hard-gelatin capsule. The aim of this prospective study is to determine the efficacy and safety of OPERA® supplementation in a series of patients affected by arthralgia during AI treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Karnofsky performance score≥70
* Indication for AI treatment in adjuvant setting for breast cancer
* Arthralgia with grade ≥0-1

Exclusion Criteria:

* Concomitant diseases, e.g. diabetes, renal insufficiency, alcohol abuse
* Concomitant rheumatological disease (Rheumatoid arthritis, Spondyloarthropathies, Psoriatic arthritis, etc.)
* Concomitant endocrinological disease (Acromegaly , Emocromatosis, etc)
* Any conditions that would complicate arthralgia assessment (e.g. Trauma, Glucocorticoid withdrawal, Hypertrophic osteoarthropathy, Osteoarthritis, Avascular necrosis, Gout, Systemic lupus erythematosus, Septic arthritis, etc.)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Reduction of AI induced arthralgia at 6 months | 6 months
  Reduction of AI-induced arthralgia assessed with VAS scale (0, no pain, to 5, worst pain)
Reduction of AI induced arthralgia at 6 months | 6 months
  Reduction of AI-induced arthralgia assessed with PRAI questionnaire (16 items that query pain severity over the last 7 days in eight joints using a rating scale of 0-10, with 10 being greatest severity)

SECONDARY OUTCOMES:
QoL | 6 months
  Quality of life assessed with FACT-ES questionnaire (19 items which assess endocrine complaints and adverse effects with response scores ranging from 0 to 4 ('not at all', 'a little bit', 'somewhat', 'quite a bit', and 'very much.')
Compliance | 6 months
  Compliance to AI therapy (percentage of patients that have not discontinued and/or changed originally prescribed anti-aromatase inhibitor)

CONTACTS AND LOCATIONS:
Overall Officials: Isacco Desideri, MD, Principal Investigator — Radiation Oncology Unit, AOU Careggi; Lorenzo Livi, MD, Study Chair — Radiation Oncology Unit, AOU Careggi
Locations (1):
- Azienda Ospedaliero Universitaria Careggi, Florence, Italy

IPD SHARING:
Plan to Share IPD: No